CLINICAL TRIAL: NCT02000726
Title: Neuroimaging Predictors of Antidepressant Treatment Outcome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding to complete the trial phase of the study.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Marta Pecina Iturbe, MD PhD, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: HUM00073082
Record Dates: First submitted 2013-10-24; First posted 2013-12-04 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo and Citalopram (Experimental): 4 weeks of 1 placebo pill/day and 12 weeks of citalopram 20-40 mg/day
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Fast acting antidepressant-like treatment. administered i.v. during the fMRI scanning session

INTERVENTIONS:
Drug: Placebo
Drug: Citalopram
  Other Names: Celexa
Drug: Fast acting antidepressant-like treatment. administered i.v. during the fMRI scanning session — Fast acting antidepressant-like treatment administered intravenously for 35 min. during the fMRI scanning session.

SUMMARY:
Current medical therapies for depression take weeks to achieve full efficacy, and are ineffective in many patients or cause intolerable side effects, emphasizing the need for a deeper understanding of depression and its treatment. Identifying early brain biomarkers of treatments responses seems necessary to improve antidepressant treatment outcome. In this study we aim to detect early brain responses to a fast acting antidepressant-like treatment administered intravenously during a Real-Time Neurofeedback functional magnetic resonance imaging (MRI) Task to predict antidepressant treatment outcome in depression. At completion of the neuroimaging task, participants will enter a placebo-controlled clinical trial with a selective serotonin reuptake inhibitor (SSRI).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will include Hamilton Depressive Rating Scale (HDRS) scores >15 and Snaith-Hamilton Pleasure Scale scores (SHAPS) > 7.

Exclusion Criteria:

suicidal ideation, comorbid conditions that are medical, neurological or psychiatric, pregnancy, use of hormones (including birth control) or use of psychotropic agents. We will only permit certain past anxiety disorder diagnoses, including generalized anxiety, panic, agoraphobia, social phobia.

We will also exclude left-handed individuals and patients who have used any centrally acting medications, nicotine, or recreational drugs within the past 2 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Blood-oxygen-level dependent (BOLD) responses during the Real-Time Neurofeedback Task. | BOLD responses will be assessed at baseline and depression severity will be assessed at baseline

SECONDARY OUTCOMES:
Depression severity assessed with several depressive questionnaires. | Every two weeks until the end of the trial (16 weeks total), or until the participants leave the study.

OTHER OUTCOMES:
Neuropsychological functioning of patients with depression | At baseline
  Affect processing: Emotional Words Task and Facial Emotion Perception test. Attention and Inhibitory Control: Parametric Go/NoGo, Trail Making test and the Stroop Color Word test .
  Inferential Reasoning (including cost-benefit analysis): Delayed Discounting of Money Rewards, Iowa Gambling Task, Common Difference effect gambling task and the WCST.
BDNF Val66Met single nucleotide polymorphism(SNP)genotyping | At baseline
  5ml of blood drawn per participants will be used for genotyping

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Ann Arbor, Michigan, United States